CLINICAL TRIAL: NCT06294392
Title: KEEP Connecting Kin: Improving Outcomes for Informal Kinship Care Families Via an In-Home Parenting and Peer-Support Program
Brief Title: KEEP Connecting Kin
Acronym: KEEP-CK
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Social Learning Center (Other)
Collaborators: Office of Planning, Research & Evaluation (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stacey Tiberio, Principal Investigator, Oregon Social Learning Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 90FA3010
Record Dates: First submitted 2024-02-14; First posted 2024-03-05 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Internalizing Behavior; Externalizing Behavior; Child Permanency; Parenting; Parent Stress; Service Utilization

STUDY DESIGN:
Intervention Model Description: Informal kinship caregivers will be randomly assigned to receive the KEEP-CK program either immediately or after waiting 10 months using a randomized blocked design. Blocking factors include: (a) the length of time that the child has been living in informal kinship care (<=6 months, 7 months to <2 years, or >=2 years); (b) child age (4 to 12 years, or 13+ years); and (c) low (or not low) resource families, defined by an annual household income below (or above) 150% of the federal poverty level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KEEP-CK (Experimental): Participants who are randomly assigned to the KEEP-CK condition will participate in 16 weekly group sessions with 8-12 other informal kinship caregivers, and receive manualized content related to positive parenting skills, and peer-to-peer supports and recommendations for services.
  Interventions: Behavioral: KEEP-CK
- "Services as usual" (SAU) waitlist control (No Intervention): Participants who are randomly assigned to the "services as usual" (SAU) waitlist control condition will be eligible to receive SAU that are available to all informal kinship caregivers in Oregon. Participants who ask about receiving supports will be referred to the Oregon Kinship Navigator, which is a statewide kinship navigator program that is available to all informal kinship caregivers in Oregon regardless of their participation in this study. Participants in the SAU waitlist control condition will be offered the opportunity to participate in a KEEP-CK group after 10 months, with these participants only contribute data to the SAU control condition for the impact analyses.

INTERVENTIONS:
Behavioral: KEEP-CK — The KEEP-CK model focuses on optimizing the role of kinship parents as the agents of positive change for children and youth. KEEP-CK groups for kinship parents are delivered by two co-group leaders for 16 weeks. Sessions are 90 minutes each week. The same group of 8-12 kinship parents attends each week. Each KEEP-CK group follows a manualized curriculum that emphasizes tailoring the content to the unique needs and cultures of the parent in the group and the youth in their care. The key parenting principles of the model include: (a) reinforce normative and prosocial behavior, (b) incentivize the behavior that parents want to promote, (c) build cooperation, (d) teach new behaviors, (e) use non-harsh effective limit setting, and (f) manage emotions while parenting. The key services connection elements of the model include: (a) parent discussions of services they are using or have used and (b) KEEP-CK group leaders share examples from a list of statewide and national services.
  Arms: KEEP-CK

SUMMARY:
The current study provides a unique opportunity to conduct a summative evaluation of the KEEP Connecting Kin (KEEP-CK) program by leveraging extant relationships with Oregon's Child Welfare System (CWS), Self-Sufficiency Program (SSP), and our community partners to address the needs of informal kinship families and the youth in their care. Specifically, a randomized "services-as-usual" (SAU) waitlist control design plus qualitative methods will be used to evaluate the immediate (post-intervention) and sustained (10 month) impacts of the KEEP-CK program on child, adult, and service utilization outcomes, and prevention of entry into the CWS.

DETAILED DESCRIPTION:
In the 2022 Oregon census, it was estimated that for every child placed in kinship foster care, there are 14 children being raised by kin outside of the child welfare system (CWS), with ~37,000 children being raised by kin and ~17,000 of those by grandparents. Kin caregivers, in particular those who are informal or voluntary, have fewer supports compared to non-relative (foster) caregivers and kin caregivers who are licensed by the CWS. Kin families are far less likely to access and utilize services in multiple systems. Thus, there is a great need to provide kin families with resources and keep youth who are living in kinship care out of the CWS.

"Keeping Parents Supported and Trained" (KEEP) was initially developed to focus on foster and kinship families involved in the CWS. In three prior NIH-funded randomized controlled trials, KEEP has shown positive impacts on youth and parent outcomes, and placement stability. KEEP has been scaled-up statewide in Oregon for CWS-involved families. The current study will focus on informal kinship care, thereby adding to an emerging body of evidence on the benefits of providing enhanced parenting and peer support to families by scaling-out the KEEP program to serve kin families outside of the CWS. This research builds on an initial study, "KEEP Connecting Kin" (KEEP-CK), where KEEP was adapted for informal kin, currently underway with participant recruitment ending in October 2023.

The proposed study (KEEP-CK#2) leverages our on-going relationships with state leadership in the CWS and SSP, and our community partners delivering KEEP-CK in Study #1 statewide in Oregon. In Study #2, a randomized "services-as-usual" (SAU) waitlist control design plus qualitative methods will be used to conduct a summative evaluation of the KEEP-CK program by recruiting N = 192 kinship families to examine the immediate (post-intervention) and sustained (10 month) impacts of the program on child, adult, and service utilization outcomes and prevention of entry into the CWS. Research questions include:

Aim 1 (impact on child and adult outcomes): The KEEP-CK program is posited to improve child and adult outcomes at the end of the intervention, and such effects are posited to be sustained at 6 months after the end of the intervention (10 months post baseline), compared to those who received SAU. Targeted child outcomes include (a) child well-being (i.e., behavioral and emotional functioning, including child internalizing and externalizing behaviors) and (b) child permanency (i.e., placement stability and permanency of placements). Targeted adult outcomes include (c) parenting practices and (d) parent/caregiver stress.

Aim 2 (impact on use of services): The KEEP-CK program is posited to increase parents' access to and use of services from multiple systems (e.g., Oregon Kinship Navigator, financial, educational, mental health, medical, legal) at post-intervention and follow-up compared to those who received SAU.

Aim 3 (impact on prevention of entry into the CWS): The KEEP-CK program is posited to reduce the likelihood that youth who are living in kinship care enter into the CWS by the 10-month follow-up assessment, compared to youth whose kinship caregivers received SAU.

Aim 4 (parent and youth perspectives): Qualitative methods will be used to evaluate families' satisfaction with and perspectives on the impact of KEEP-CK on child and adult outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Informal kinship caregivers in Oregon are defined as relatives or fictive kin who are caring for children between the ages of 4 to 18 years outside of the child welfare system with no birth/step parent living in the home.

Exclusion Criteria:

* Informal kinship caregivers in Oregon who have previously participated in a KEEP or KEEP-CK group, or have a partner living in their home who has previously participated in a KEEP or KEEP-CK group.
* Focal child is not between the ages of 4-18 years at the baseline assessment.
* Focal child has been adopted by the kinship parent at the baseline assessment.
* Focal child is not living with the kinship caregiver full time (e.g., babysitting/weekends/vacations) at the baseline assessment.
* Focal child is in child welfare at the baseline assessment.
* Focal child is living with the kinship caregiver in a certified foster home at the baseline assessment.
* Focal child has a developmental disability or delay that impairs their ability to be responsive to the parenting content of KEEP-CK.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 192 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Mean change in youth well-being (i.e., behavioral and emotional functioning, including child internalizing and externalizing behaviors) | Baseline, and 4- and 10-months post-baseline
  Youth well-being will be measured via kinship parent report using the Child Behavior Checklist (CBCL) at baseline and 4- and 10-months post-baseline. The CBCL has eight subscales (anxious/depressed, withdrawn/depressed, somatic complaints, social problems, thought problems, attention problems, rule-breaking behavior [delinquency], and aggressive behavior), which make up three broadband scales: total behavior, internalizing, and externalizing problems.
Mean change in child permanency (i.e., placement stability and permanency of placements) | Baseline, and 4- and 10-months post-baseline
  All children will be living in informal kinship care at the time of the baseline assessment. Changes in the child's placement setting (living conditions) will be measured via kinship parent report using the Change of Placement questionnaire at 4- and 10-months post-baseline.
Mean change in parenting practices and parent/caregiver stress. | Baseline, and 4- and 10-months post-baseline
  Parenting practices and parent/caregiver stress will be measured via the Parent Daily Report (PDR) at baseline and 4- and 10-months post-baseline. The PDR assesses whether the parent found any of the focal child's internalizing and externalizing behaviors to be stressful, and the types of positive reinforcement and discipline that were used with the child.
Mean change in parent/caregiver stress. | Baseline, and 4- and 10-months post-baseline
  Parent/caregiver stress will be measured via a shortened version of the Parenting Stress Index (PSI) short form at baseline and 4- and 10-months post-baseline to assess two domains, including parental distress, and parent-child dysfunctional interaction.
Mean change in parenting practices. | Baseline, and 4- and 10-months post-baseline
  Parenting practices will be measured via the Alabama Parenting Questionnaire (APQ) short form at baseline and 4- and 10-months post-baseline. The APQ short form assesses positive parenting, and the types of, and consistency with which, discipline was used with the focal child.
Mean change in parents' use of services from multiple systems (financial, educational, mental health, medical, legal) | Baseline, and 4- and 10-months post-baseline
  Parents will complete the Service Utilization Survey (SUS) at baseline and 4- and 10-months post-baseline, which is a measure of need for, and use of, health care and social services. Parents report on services that they have sought and used for themselves or the focus child over a 4- to 6-month period. The types of services include: housing, legal matters, financial, parenting support, medical, counseling/mental health, education, extracurricular activities, and social support from friends/relatives.

CONTACTS AND LOCATIONS:
Overall Officials: Stacey Tiberio, Ph.D., Principal Investigator — Oregon Social Learning Center
Locations (1):
- Oregon Center Learning Center, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT06294392/SAP_000.pdf